CLINICAL TRIAL: NCT00307827
Title: A Phase 2, Randomized, Double-blind, Multicenter, Dose-exploration Study of Visilizumab in Subjects With Intravenous Steroid-refractory Ulcerative Colitis
Brief Title: Study of Visilizumab in Subjects With Intravenous Steroid-Refractory Ulcerative Colitis (IVSR-UC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Canceled
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 291-418; 2005-003482-17 (EudraCT Number)
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Ulcerative Colitis
Keywords: Steroid-Refractory; IVSR-UC; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — visilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Visilizumab low dose level
  Interventions: Drug: Visilizumab
- Arm 2 (Experimental): Visilizumab middle dose level
  Interventions: Drug: Visilizumab
- Arm 3 (Experimental): Visilizumab high dose level
  Interventions: Drug: Visilizumab

INTERVENTIONS:
Drug: Visilizumab — Visilizumab administered intravenously once per day for two days
  Other Names: Nuvion®; HuM291

SUMMARY:
The purpose of this study is to assess the efficacy, immunogenicity, and safety of various doses of visilizumab in subjects with intravenous steroid-refractory ulcerative colitis (IVSR-UC) and to evaluate optimal dosing.

DETAILED DESCRIPTION:
PDL BioPharma, Inc. was formerly known as Protein Design Labs, Inc.

ELIGIBILITY:
Inclusion Criteria

Eligible subjects will be considered for inclusion in this study if they meet all of the following criteria:

* Males and females, 18 years of age or older.
* Diagnosis of ulcerative colitis (UC), as verified by endoscopy performed within 60 months prior to consent.
* Severe active disease, as defined by modified Truelove Witts severity index (MTWSI) >= 11 at consent, with a confirmatory MTWSI >= 10 on or after the fifth consecutive day of intravenous (IV) steroids and within 1 day prior to randomization.
* Mayo score >= 10 and Mayo mucosal subscore >= 2 after a minimum of 3 consecutive days (ie, on or after the fourth consecutive day) of IV steroids.
* Adequate contraception from the day of consent through 3 months after the last dose of study drug.
* Negative serum pregnancy test at screening.
* Negative Clostridium difficile test within 10 days prior to randomization.
* Signed and dated informed consent and Health Insurance Portability and Accountability Act (HIPAA) if applicable.

Exclusion Criteria

Subjects will be ineligible for this study if they meet any one of the following criteria:

* UC requiring immediate intervention.
* History of total proctocolectomy, or subtotal colectomy with ileorectal anastomosis
* Presence of ileostomy.
* White blood cell count less than 2.5 x 10^3/mcL; platelet count less than 150 x 10^3/mcL; or hemoglobin level less than 8 g/dL.
* Active medically significant infections, particularly those of viral etiology, eg, known cytomegalovirus (CMV) colitis. This includes any incidence of medically significant opportunistic infections within the past 12 months.
* Live vaccination within 6 weeks prior to randomization.
* Significant organ dysfunction, including cardiac, renal, liver, central nervous system (CNS), pulmonary, vascular, gastrointestinal, endocrine, or laboratory abnormality.
* History or treatment of lymphoproliferative disorder (LPD) or malignancy within the past 5 years (excluding nonmelanoma skin cancer or carcinoma in situ of the cervix).
* Seropositivity for infection with human immunodeficiency virus (HIV-1), hepatitis B virus (HBV) surface antigen, or hepatitis C virus (HCV).
* Pregnancy or nursing.
* Treatment with a first dose of infliximab or another anti-TNF-a drug within 4 weeks of randomization, or treatment with a subsequent dose of an anti-TNF-a drug within 2 weeks of randomization.
* Treatment with cyclosporine or tacrolimus (FK506) within 2 weeks prior to randomization.
* Treatment with any other investigational drugs or therapies within 60 days prior to randomization, except those mentioned in the two exclusion criteria above.
* Unwilling or unable to discontinue all UC drugs, except glucocorticoids and oral 5-ASA, immediately prior to randomization.
* Nontherapeutic levels of chronic antiseizure medications in subjects with a prior history of seizures.
* Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each of the three visilizumab dose groups who respond to treatment in the dose-exploration portion of this study (Stage 1). | Day 45

SECONDARY OUTCOMES:
Comparison of subjects in the three visilizumab dose groups | During the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — Abbott
Locations (16):
- United States (5):
  - Site Reference ID/Investigator# 71894, Savannah, Georgia
  - Site Reference ID/Investigator# 71897, Worcester, Massachusetts
  - Site Reference ID/Investigator# 71913, Manhasset, New York
  - Site Reference ID/Investigator# 71895, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 71896, Cleveland, Ohio
- Canada (2):
  - Site Reference ID/Investigator# 71875, Hamilton
  - Site Reference ID/Investigator# 71873, Winnipeg
- Croatia (2):
  - Site Reference ID/Investigator# 72338, Osijek
  - Site Reference ID/Investigator# 72334, Zagreb
- Site Reference ID/Investigator# 72345, Bologna, Italy
- Russia (4):
  - Site Reference ID/Investigator# 72314, Moscow
  - Site Reference ID/Investigator# 71953, Nizhny Novgorod
  - Site Reference ID/Investigator# 72315, Saint Petersburg
  - Site Reference ID/Investigator# 72342, Saint Petersburg
- Spain (2):
  - Site Reference ID/Investigator# 72368, Badalona - Barcelona
  - Site Reference ID/Investigator# 72366, Majadahonda (Madrid)